CLINICAL TRIAL: NCT04946981
Title: A Placebo Controlled, Randomised, Crossover Clinical Trial to Evaluate the Effect of Turmipure Gold® in Muscle Pain and Function Recovery in Moderately Active Adults
Brief Title: Recovery and Muscle Function After Supplementation With Turmeric
Acronym: RECOFAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Givaudan France Naturals (Industry)
Collaborators: Atlantia Food Clinical Trials (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AFCRO-128
Record Dates: First submitted 2021-06-21; First posted 2021-07-01 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Muscle Soreness; Pain; Muscle Damage
Keywords: Turmeric; Curcuminoids; Sport performance & recovery
MeSH Terms: conditions — Myalgia; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Randomized Crossover_Sequence 1 (Other): Participants who meet the eligibility criteria will be randomized and will receive first the experimental product Turmipure GOLD® during the first study phase and then the placebo control during the second study phase. Both study phases are separated by a washout period of minimum 14 days.
  Interventions: Dietary Supplement: Turmipure Gold®; Dietary Supplement: Placebo
- Randomized Crossover_Sequence 2 (Other): Participants who meet the eligibility criteria will be randomized and will receive first the placebo control during the first study phase and then the experimental product Turmipure GOLD® during the second study phase. Both study phases are separated by a washout period of minimum 14 days.
  Interventions: Dietary Supplement: Turmipure Gold®; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Turmipure Gold® — TPG: Turmipure GOLD® - 1 capsule per day - as prescribed
Dietary Supplement: Placebo — Placebo: colored acacia gum - 1 capsule per day - as prescribed

SUMMARY:
The objective of the study is to test the capacity of a five-day supplementation of Turmipure Gold® to improve exercise-induced muscle pain and function recovery in moderately active adults after exercise-induced muscle damage

ELIGIBILITY:
Inclusion Criteria:

* Healthy free-living males
* Age: 25-45 years old
* Have a BMI between 18.5 and 28 kg/m²
* Moderately active with running 15-20 km per week
* With 1 to 4h of training per week, with maximum 1h of lower body heavy-load or resistance training (e.g., Hill running or hiking, HIT exercise, Squats, Lunges, Leg-press, Bench steps, etc.)
* Consent to the study protocol and to comply with study product
* Willing to limit caffeine, smoking, and alcohol consumption during the entire study period with no more than 5 cigarettes per day and 2 drinks. Also, alcohol consumption will not be allowed 24hours prior to exercise-induced muscular damage
* Willing to refrain from training for 3 days before the first test, 5 days before each damage-inducing exercise and during each supplementation phase, including active recovery exercises such as swimming, cycling at low intensity, unusual distance walking (however such should be encouraged during the 14 days wash-out)
* Willing to refrain the use of anti-inflammatory/pain reliever drugs such as paracetamol, NSAIDs, etc., during each supplementation phase, from 24 hours prior to 72 hours following the exercise-induced muscular damage
* Willing to refrain from 'recovery' treatments over the 72 hours following the damage inducing exercise such as:

  1. Hydrotherapy - cold water immersion, hot water immersion, or contrast therapy (as well as Jacuzzis, Steam baths, or Saunas)
  2. Massage - self, foam rolling, etc.
  3. Stretching
  4. Compression garments
  5. Topical applications - Tiger Balm, Deep Heat etc.

Exclusion Criteria:

* Participants with any indicators of arthritis, joint disorders chronic pain syndrome, muscle disorder diseases (e.g., fibromyalgia, etc.)
* History of surgery or significant injury in joints or in the lower limb in the last six months prior to study enrolment, or an anticipated need for surgical or invasive procedure that will be performed during the study
* Using omega-3-fatty acid, probiotic supplements, vitamins, minerals, or any dietary supplements (including botanicals), especially to maintain joint health 4 weeks prior to screening and during the entire study. Potential supplements include but are not limited to Beta-alanine, Creatine, HMB, Carnosine, Taurine, androstenedione, DHEA, Whey protein, or a pre-workout supplement
* Following any specific diet such as high-protein, vegetarian, vegan, etc
* Taking any drugs such as antibiotics, laxatives, or immunosuppressant drugs
* History of glucocorticoid injection or hyaluronic acid injections within 3 months prior to enrolment
* Participants near or in the peak of training for an athletic race (half or marathon, cycling tour or triathlon)
* History or current significant cardiovascular, pulmonary, renal, liver, digestive (including an inflammatory bowel disease), infectious disease, systemic disease, immune disorder, or metabolic/endocrine disorders (including diabetes mellitus) or other disease that would preclude supplement ingestion and/or assessment of study objectives, including uncontrolled hypertension, uncontrolled thyroidism or lipidaemia that is not on stable medication for at least 3 months.
* Participant has any concurrent medical or psychiatric condition that, in the opinion of the Investigator, would compromise his/her ability to comply with the study requirements
* Participant with history of drug and / or alcohol abuse at the time of enrolment
* Any previous or current cancer diagnosis (including a benign or malign tumour of intestine or colon)
* Current illnesses which could interfere with the study (e.g., prolonged severe diarrhoea, regurgitation/severe, difficulty swallowing)
* Known allergy to components of the test product or sensitivity to herbal products or with a medical history of food allergies
* Participants taking any anticoagulant or heparin treatment (including aspirin)
* Clinically significant abnormal laboratory results at screening
* Participant currently involved in any other clinical trial or having participated in a trial within 90 days prior to randomisation.
* Any other condition which in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject.
* History of non-compliance with medical treatments or recommendations.
* Participants who are required to perform squatting motions or descend a lot of stairs in their daily work activities, which may be painful following the Exercise Induced Muscle Damage.

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Change on Perceived Muscle Soreness | 72 hours
  Perceived Muscle Soreness in quadriceps during squatting activities assessed by VAS (0-100 mm, after two tries)

SECONDARY OUTCOMES:
Change on Muscle damage | 72 hours
  Muscle damage assessed by circulating levels of Creatine kinase in blood samples
Change on Isometric Muscle function recovery | 72 hours
  Muscle function recovery assessed on quadriceps muscular function during isometric contractions recording the torque (Nm) using Biodex
Change on Isokinetic Muscle function recovery | 72 hours
  Muscle function recovery assessed on quadriceps muscular function during isokinetic extensions recording the torque (Nm) using Biodex
Change on Muscle power recovery | 72 hours
  Muscle power recovery assessed by Peak power (Watts) using vertical jump tests (best performance and average of 3 tries)
Change on Muscle ROM recovery | 72 hours
  Muscle ROM recovery assessed by Range Of Movement using a goniometer (knee flexion)
Change on Perceived wellness and well-being | 72 hours
  Perceived wellness and well-being is assessed by a psychometric test evaluating fatigue, sleep quality, general muscle soreness, stress, and mood (0-25, 25 indicating best feelings of wellness and well-being)
Change on Perceived exertion during exercise | 30 min
  Perceived exertion through breathing difficulty during exercise assessed by the Borg Rating of Perceived Exertion (0-10, 10 indicating maximal difficulty)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Dinan, Professor, Principal Investigator — Atlantia Food Clinical Trials; Trevor Wood, PhD, Principal Investigator — Sport Physiologist University College Cork
Locations (1):
- Atlantia Food Clinical Trials, Cork, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Schonenberger KA, Laval J, Woods T, Truillet R, Naranjo-Modad S, Mettler S, Fanca-Berthon P. A randomized, placebo-controlled, crossover clinical trial to evaluate the effect of a turmeric formulation on muscle soreness and function recovery in moderately active adults. J Int Soc Sports Nutr. 2025 Dec;22(1):2568048. doi: 10.1080/15502783.2025.2568048. Epub 2025 Oct 3. PMID 41040018